CLINICAL TRIAL: NCT01189461
Title: An Open Label, One Year, Non-Comparative Study To Evaluate The Safety And Tolerability Of Intravitreous Pegaptanib Sodium In Patients With Diabetic Macular Edema
Brief Title: Study To Evaluate Safety And Tolerability Of Pegaptanib Sodium In Patients With Diabetic Macular Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5751036
Record Dates: First submitted 2010-07-23; First posted 2010-08-26 (Estimated); Results first posted 2013-09-06 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-06

CONDITIONS: Anti- VGF Inhibitor; Diabetic Macular Edema; Diabetic Retinopathy
Keywords: pegaptanib sodium; diabetic macular edema
MeSH Terms: conditions — Diabetic Retinopathy | interventions — pegaptanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pegaptanib sodium arm (Experimental): all patients will receive pegaptanib sodium
  Interventions: Drug: pegaptanib sodium

INTERVENTIONS:
Drug: pegaptanib sodium — Upon enrollment, all subjects will be treated in the study eye with pegaptanib sodium 0.3 mg at the investigators' discretion based on visual acuity assessment up to a maximum of 48 weeks. The minimum dosing interval between injections will be at least 6 weeks.

SUMMARY:
This study will asses sthe safety of pegaptanib sodium in patients with diabetic macular edema. The hypothesis is that pegaptanib is safe and efficacious in patients with diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Subjects with documented clinical diagnosis of diabetic macular edema (DME) with proliferative or non proliferative diabetic retinopathy.
* Subjects, who according to the clinical assessment of the investigator, may benefit from anti-VEGF therapy including those subjects who were participating in the A5751013 study and who, in the investigator's opinion, may benefit from continued pegaptanib sodium therapy.

Exclusion Criteria:

* Eyes with prior scatter (panretinal) photocoagulation within 4 months prior to baseline or anticipated scatter (panretinal) photocoagulation within the next 6 months.
* Presence of any abnormality that is likely to confound assessment of visual acuity improvement in eyes in which macular edema resolves, or improves, such as non-perfusion for >1 disc area involving the foveal avascular zone (FAZ - involving 2 or more quadrants centered around the foveal avascular zone), epiretinal membrane associated with signs of contraction and/or significant opacification (i.e. striae within 1 disc diameter of the foveal center), or presence of chorioretinal atrophy involving the center of the macula.
* Vitreomacular traction determined clinically and/or by optical coherence tomography (OCT), which, in the investigator's opinion, contributes to the macular edema (or causes associated foveal detachment), and would preclude improvement with pegaptanib sodium.
* Any other cause of macular edema such as vitreous extension, or entrapment to anterior segment wound, or any retinal vein occlusion involving the macula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- Finland (2):
  - Kuopion Yliopistollinen sairaala, Kuopio
  - PHSOTEY / Silmätautien klinikka, Lahti
- Spain (6):
  - Hospital Naval Del Ferrol, Ferrol, A Coruña
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona, Girona
  - Hospital Ntra. Sra. de La Esperanza, Santiago de Compostela, La Coruña
  - Hospital Universitario Clinico San Carlos, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
- Sweden (2):
  - Stockholms Ogonklinik, Stockholm
  - Ogonkliniken, Centrallasarettet, Västerås
- United Kingdom (2):
  - Frimley Park Hospital, Frimley, Camberley, Surrey
  - Kings College Hospital, London

REFERENCES:
- [Derived] Sivaprasad S, Browning RC, Starita C. An open-label, one-year, noncomparative study to evaluate the safety and tolerability of intravitreal pegaptanib sodium in patients with diabetic macular edema. Clin Ophthalmol. 2014 Aug 21;8:1565-71. doi: 10.2147/OPTH.S68498. eCollection 2014. PMID 25187694
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5751036&StudyName=Study%20To%20Evaluate%20Safety%20And%20Tolerability%20Of%20Pegaptanib%20Sodium%20In%20Patients%20With%20Diabetic%20Macular%20Edema

RESULTS

PARTICIPANT FLOW:
Groups:
- Macugen: Macugen (pegaptanib sodium) 0.3 milligram (mg) intravitreal injection administered once every 6 weeks into the study eye up to Week 48.
Period: Overall Study
Arm/Group | Macugen
Started | 46
Completed | 12
Not Completed | 34
Not completed — Lack of Efficacy | 13
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 6
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 2
Not completed — Did not meet entrance criteria | 3
Not completed — Other | 8

BASELINE CHARACTERISTICS:
Arm/Group | Macugen
Number analyzed (Participants) | 46
Age Continuous [Mean (Standard Deviation); unit: years] | 65.0 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Ocular and Non-Ocular Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Total number of participants who had ocular and non-ocular AEs was reported.
Time Frame: Baseline up to 30 days after last dose
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication. Same participant may be represented in more than 1 category.
Measure: Number; unit: participants
Arm/Group | Macugen
Number analyzed (Participants) | 46
participants
  Ocular AEs | 10
  Non-ocular AEs | 8

2. Secondary Outcome: Incidence of Ocular and Non-Ocular Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Total number of participants who had ocular and non-ocular SAEs was reported.
Time Frame: Baseline up to 30 days after last dose
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Macugen
Number analyzed (Participants) | 46
participants
  Ocular SAEs | 0
  Non-ocular SAEs | 3

3. Primary Outcome: Mean Total Number of Injections
Description: Mean number of injections per participant was calculated as (number of injection administered per participant - 1)/duration of treatment. Mean number of injections administered for total participants was summarized.
Time Frame: Baseline up to Week 48 (End of treatment)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | Macugen
Number analyzed (Participants) | 46
injections | 3.24 (1.037)

4. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Score at Week 48 (End of Treatment)
Description: VA indicated sharpness or clarity of vision. BCVA assessed by early treatment diabetic retinopathy study chart using 4 meter (m), 1m distance, or if participant was able to count fingers, perceive hand motion or light. At 4m (>= 20 letters), VA score=number of letters correct plus 30 (credited for 30 letters at 1m); otherwise , VA score=number of letters read correctly at 1m plus number read at 4m (if any). If no letters were read correctly at 4m or 1m, VA score= 0, which were excluded from summary statistics calculation. BVCA score ranged: 0 (poor eyesight) to 78 (best eyesight).
Time Frame: Baseline, Week 48 (End of treatment)
Population: Full analysis set included all enrolled participants who received at least 1 dose of study medication. Here 'N' (number of participants analyzed) signifies participants who had BVCA score greater than 0 at baseline and 'n' signifies those who were evaluable at each specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Macugen
Number analyzed (Participants) | 42
units on a scale
  Baseline (n= 42) | 58.93 (16.468)
  Change at Week 48 (n= 14) | 2.21 (7.536)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Macugen
Serious Adverse Events (participants affected / at risk) | 3/46
Other Adverse Events (participants affected / at risk) | 16/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macugen (N=46)
Myocardial infarction (Cardiac disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macugen (N=46)
Anaemia (Blood and lymphatic system disorders) | 1
Cataract (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Conjunctival hyperaemia (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Eye discharge (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Macular oedema (Eye disorders) | 3
Maculopathy (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 2
Vitreous floaters (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastric polyps (Gastrointestinal disorders) | 1
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Biopsy vocal cord (Investigations) | 1
Carcinoembryonic antigen increased (Investigations) | 1
Intraocular pressure increased (Investigations) | 1
Headache (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.